CLINICAL TRIAL: NCT05004168
Title: The Efficacy of Sun Protection Factor (SPF) Against UV-B and UV-A of Cosmetic Products
Brief Title: Sun Protection Factor (SPF) / UVA Protection Factor Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Collaborators: PT Paragon Technology and Innovation (Unknown)
Responsible Party: Principal Investigator, Prof. dr. Franciscus D. Suyatna, PhD, SpFK, Clinical Pharmacology Professor, Indonesia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CRSU.P.SPF_Paragon/02.20/07.03
Record Dates: First submitted 2021-07-08; First posted 2021-08-13 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Sunscreen Agents
Keywords: Sun Protection Factor; Sunscreen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SPF evaluation (Experimental): Healthy male or female subjects with Fitzpatrick Skin Type of II-IV were included in the SPF study
  Interventions: Other: Day Gel-0120; Other: P5 Reference Standard (SPF 35 reference)

INTERVENTIONS:
Other: Day Gel-0120 — Two milligrams of test article applied to the test area. The test products are Day Gel-0120C and Day Gel-0120-D. The products are applied together on the test area with
Other: P5 Reference Standard (SPF 35 reference) — The reference product is P5 according to ISO 24444:2019. The application of reference product is similar with test product.

SUMMARY:
Evaluation of the effectiveness of sunscreen products by determining its Sun Protection Factor (SPF) against UV-B and UV-A

DETAILED DESCRIPTION:
Sunscreen is intended to protect the skin from sun burn but since the amount of protection needed varies among individuals, sunscreen manufactures offer consumers difference levels of protection. These different levels of protection are expressed as a numerical value called the sun protection factor or SPF. The SPF is the ratio between the minimal erythema dose (MED) of sunscreen product of the protected skin and the MED of the unprotected skin. The minimal erythema dose in human skin is defined as the lowest ultraviolet B (UV-B) dose produces the first perceptible unambigous erythema with defined border appearing over most of the field of UVB exposure 16 - 24 hours after UVB exposure.

The UVA protection factor is the ratio between the Minimal Persistent Pigmentation Darkening Dose (MPPDD) of sunscreen product of the protected skin and the MPPDD of the unprotected skin. The threshold response will be taken as an unequivocal pigment darkening with distinct border which persisted for at least 2 hours.

The test products are Day Gel-0120-C and Day Gel-0120-D with active ingredients ethylhexyl methoxycinnamate, Diethylamino hydroxybenzoyl hexyl benzoate

ELIGIBILITY:
Inclusion criteria:

1. Healthy male or female, 18-60 years of age
2. Fair skin with skin type II-IV of Fitzpatrick's skin type
3. Able to understand and comply to the investigators instruction.
4. Able to read, understand and sign up informed consent form.

Exclusion criteria:

1. Subject with a history of abnormal response to sunlight or those taking medication which might produce an abnormal response to sunlight
2. Subject exhibiting current sun burn, sun tan, uneven skin tone, or visible skin disease which might be confused with a reaction from the test material or which might interfere with evaluation of test results
3. Individuals who are under doctor's care
4. Female subjects who indicate that they are pregnant or nursing
5. Individuals with known hypersensitivity to any sunscreen products
6. Individuals accustomed to using tanning beds

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2020-09-24 (Actual); Study Completion 2020-09-24 (Actual)

PRIMARY OUTCOMES:
To measure the SPF Value of the teat product | 2-24 hours post exposure
  The mean of SPF value from all the subject

CONTACTS AND LOCATIONS:
Overall Officials: Frans Suyatna, Prof, PhD, Principal Investigator — Clinical Research Supporting Unit, Faculty of Medicine, University of Indonesia
Locations (1):
- Clinical Research Supporting Unit, Jakarta Pusat, DKI Jakarta, Indonesia

REFERENCES:
- [Background] Heckman CJ, Chandler R, Kloss JD, Benson A, Rooney D, Munshi T, Darlow SD, Perlis C, Manne SL, Oslin DW. Minimal Erythema Dose (MED) testing. J Vis Exp. 2013 May 28;(75):e50175. doi: 10.3791/50175. PMID 23748556
- [Background] Donglikar MM, Deore SL. Sunscreens: A review. Pharmacognosy Journals. 2016;8(3):171-179
- See also: ISO 24444:2019-Sun Protection test methods-in vivo determination of the Sun Protection Factor (SPF) — https://www.iso.org/standard/72250.html
- See also: Sun protection test methods-In vivo determination of sunscreen UVA protection — https://www.iso.org/standard/46521.html